CLINICAL TRIAL: NCT04024189
Title: Audit of Informed Consent of Patients Undergoing Surgery
Brief Title: Patient Experience of Consent for Cancer Surgery in Light of Recent Changes to UK Law- a Questionnaire Study
Status: Completed | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 18/2117
Record Dates: First submitted 2019-06-14; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Patients were given a questionnaire/survey to complete in respect of their satisfaction of the consent process for their surgical procedure

SUMMARY:
Since the 2015 Montgomery vs Lanarkshire Health Board ruling, the consent process in the UK has had to change. In practice, this means that doctors must ask themselves whether the patient knows about the material risks of the treatment being proposed, alternatives to the treatment, and whether reasonable care has been taken to ensure the patient actually knows this. This study aims to determine patients' perspectives of consent for major cancer surgery in light of the Lanarkshire ruling.

DETAILED DESCRIPTION:
A patient satisfaction survey was administered to patients who had undergone urological, gynaecological, colorectal, and plastic surgical procedures at a specialised cancer centre where changes to consent processes in light of the Lanarkshire ruling had been implemented.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been admitted and undergone surgery within a 6 week period between April - June 2018.

Exclusion Criteria:

* Any patient who could not complete the survey questionnaire i.e. English was not their first language or to unwell to complete.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery during a 6 week period at The Christie NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Patients understanding of the risks associated with the procedure they will be having and the alternatives available to them was assessed using a study specific questionnaire. | 6 weeks
  Was the patient made aware by the clinical care team of the risks associated with their procedure and the alternatives available to them. Were they able to make an informed choice. This will be measured using a patient questionnaire
Patients views and feelings regarding their experiences in relation to support from healthcare professionals was assessed using a study specific patient questionnaire. | 6 week
  Did patients feel that healthcare professionals provided them with sufficient information and support to make an informed decision in respect of their procedure. This will be measured using a questionnaire completed by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Aziz, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.